CLINICAL TRIAL: NCT06447415
Title: Safety, Tolerability, and Preliminary Efficacy of HRS-7450 Injection in the Treatment of Acute Ischemic Stroke: a Multi-center, Randomized, Double-blind, Double-dummy, Placebo-controlled, Single Dose Incremental Phase Ib Clinical Trial
Brief Title: Safety, Tolerability, and Preliminary Efficacy of HRS-7450 Injection in the Treatment of Acute Ischemic Stroke: a Multi-center, Randomized, Double-blind, Double-dummy, Placebo-controlled Clinical Trial
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fujian Shengdi Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HRS-7450-102
Record Dates: First submitted 2024-06-03; First posted 2024-06-07 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Multi-center, randomized, double-blind and double simulated, placebo controlled, single dose escalation
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HRS-7450 (Experimental)
  Interventions: Drug: HRS-7450
- 0.9% sodium chloride injection (Placebo Comparator)
  Interventions: Drug: 0.9% sodium chloride injection

INTERVENTIONS:
Drug: HRS-7450 — HRS-7450 Injection
  Arms: HRS-7450
Drug: 0.9% sodium chloride injection — 0.9% sodium chloride injection
  Arms: 0.9% sodium chloride injection

SUMMARY:
This study is a multi-center, randomized, double-blind, double-dummy, placebo-controlled, single dose escalation study aimed at evaluating the overall safety, tolerability, and preliminary efficacy of HRS-7450 in patients with acute ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

1. Fully understand and voluntarily participate in this study, and sign an informed consent form (the informed consent form can be voluntarily signed by the individual or legal representative);
2. 18 ≤ Age ≤ 80 years old;
3. The onset time is within 4.5 to 24 hours, and medication can be completed within 24 hours of onset (onset time is defined as the patient's last normal time);
4. Clinically diagnosed as acute ischemic stroke (diagnosis follows the Chinese Guidelines for the Diagnosis and Treatment of Acute Ischemic Stroke 2023);
5. mRS score ≤ 2 before the first episode;
6. When screening, the National Institutes of Health Stroke Scale (NIHSS) scores from 3 to 25 (including both ends);
7. Female and male participants with fertility must agree to use efficient contraception measures from the signing of the informed consent form until one month after the last administration of the investigational drug, without a birth plan, and without donating sperm/eggs. (See "Contraceptive methods" in the attachment for details).

Exclusion Criteria:

1. Treatment with ateplase, teneplase, or other thrombolytic drugs;
2. Proposed endovascular treatment;
3. Intracranial hemorrhagic diseases;
4. Aortic arch dissection;
5. NIHSS awareness score 1a>2 points;
6. Epileptic seizures or neurological dysfunction after seizures, or combined with other neurological/psychiatric disorders leading to uncooperative or non cooperative physical examinations;
7. Non enhanced CT shows a low-density shadow greater than one-third of the blood supply area of the middle cerebral artery or an ASPECT score of less than 6 points in the anterior circulation;
8. Previous history of intracranial hemorrhage;
9. Intracranial tumors, arteriovenous malformations, and giant aneurysms;
10. Acute occlusion of the internal carotid artery due to carotid artery dissection;
11. Multiple infarcts in areas supplied by multiple large blood vessels;
12. Have a history of ischemic stroke, severe traumatic brain injury, or intracranial or spinal surgery in the past month;
13. Gastrointestinal or urinary system bleeding within the past 2 weeks;
14. Major surgical procedures or severe injuries within the past 2 weeks;
15. Arterial puncture that is difficult to compress and stop bleeding within the past week;
16. Active visceral bleeding;
17. After actively reducing blood pressure, systolic blood pressure ≥ 180mmHg and/or diastolic blood pressure ≥ 100mmHg;
18. Screening period examination: Blood glucose<2.8 or>22.2mmol/L, platelet<100 * 109/L, other findings suggestive of a high risk of bleeding;
19. Within the past 3 months, acute ST segment elevation myocardial infarction (MI) and/or acute decompensated heart failure occurred, and/or QTc>520 milliseconds, and/or due to acute coronary syndrome MI、 Hospitalization or involuntary coronary intervention for cardiac arrest; Or New York Heart Association Grade III/IV heart failure; Or known to have ventricular tachycardia;
20. History of severe liver disease, or aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) and/or glutamyltransferase (GGT) ≥ 3 x ULN and/or total bilirubin (TBIL) ≥ 2 x ULN.
21. Severe kidney disease with clinical significance, or eGFR<45mL/min/1.73 m2;
22. Subjects with known potential bleeding constitution or coagulation dysfunction;
23. Subjects with a known history of glucose-6-phosphate dehydrogenase deficiency or a family history;
24. Known to be allergic to any component of HRS-7450 or its formulations or placebo;
25. Received therapeutic or prophylactic doses of heparin treatment within 24 hours;
26. Oral coumarin anticoagulants with an international standardized ratio INR>2.7;
27. Use thrombin inhibitors, Xa factor inhibitors, or other anticoagulant drugs under study within48 hours;
28. Use platelet IIb/IIIa receptor inhibitors within 48 hours;
29. Pregnant women, or women of childbearing age who test positive for pregnancy, or those who are breastfeeding;
30. Participate in clinical studies of other drugs or devices within the first three months of the screening period (sign an informed consent form and receive treatment with the trial drug/device);
31. The terminal state of the disease, with an expected survival period of no more than 1 year;
32. Other situations where the researcher deems it inappropriate to participate in this experiment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2024-08-06 (Actual); Primary Completion 2025-03-18 (Actual); Study Completion 2025-06-11 (Actual)

PRIMARY OUTCOMES:
Symptomatic Intracranial Hemorrhage within 36 hours after the start of administration, The incidence of sICH | within 36 hours after the start of administration

SECONDARY OUTCOMES:
7 day mortality rate after administration | within 7days after the start of administration
The incidence of sICH 7 days after administration | within 7days after the start of administration
The incidence of ICH 7 days after administration | within 7days after the start of administration
The incidence of systemic bleeding 7 days after administration | within 7days after the start of administration
Effective reperfusion rate measured by 24-hour PWI or CTP | within 24 hours after the start of administration
24-hour MRA or CTA measurement of vascular reperfusion rate | within 24 hours after the start of administration
Infarct core volume measured by CT or MRI at 5-7 days | within 5-7days after the start of administration
24-hour NIHSS score change | within 24 hours after the start of administration
24-hour good response rate (NIHSS score reduction greater than 8 points, or NIHSS score 0-1) | within 24 hours after the start of administration
7 day NIHSS score change | within 7days after the start of administration
7 day good response rate (NIHSS score reduction greater than 8 points, or NIHSS score 0-1) | within 7days after the start of administration

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Sun Yat sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided